CLINICAL TRIAL: NCT00094354
Title: A Qualitative Study for the Development of an Intervention Among HIV-Positive Former Plasma Donors (FPDs) in Fuyang, Anhui Province, China
Brief Title: HIV Assessment in Fuyang, Anhui Province, China
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Rona Siskind, DAIDS
Other Study IDs: CIPRA CH 002A; CIPRA; Project 2
Record Dates: First submitted 2004-10-16; First posted 2004-10-18 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: HIV infected former Plasma Donors; Needs assessment; HIV-related stigma and discrimination; In-depth interview; Focus Groups
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: HIV-infected FPDs
- 2: Family members of HIV-infected FPDs
- 3: Local healthcare workers
- 4: Villagers not related to an HIV-infected individual

SUMMARY:
The purpose of this study was to examine the needs, concerns, stigmas, and social networks of HIV infected former plasma donors (FPDs) and their relatives in Fuyang, Anhui Province, China. Interviews and focus groups were used to collect data in preparation for a future, larger behavioral study for HIV infected individuals in China.

DETAILED DESCRIPTION:
The HIV epidemic in China has reached a phase of exponential growth. Among the infected are former commercial plasma donors (FPDs) in rural communities, who became infected through contaminated blood collection equipment. This study examined the needs, concerns, stigmas, social networks, and discrimination among HIV infected FPDs and their families. The study was designed to provide preliminary information and help prepare for the implementation of a second study, which evaluated community based intervention on quality of life of HIV infection villagers and HIV-related stigma.

Four groups of people were enrolled in this study: HIV infected FPDs; family members of HIV infected FPDs; local healthcare workers; and other villagers not related to an HIV infected individual. Participants were recruited based on sampling framework which stratified potential participants by gender, age, and place of residence. Selected study participants from all four groups had in-depth, one-on-one interviews approximately 2 to 3 hours in length. The interviews were taped and transcribed, and the transcriptions were coded with respect to responses. In addition, there were 2 separate focus groups; one for local healthcare workers and a second for other villagers not related to an HIV infected individual.

Information was collected from 111 participants through face-to-face, in-depth interviews (FFI) and focus group discussions (FGD). FFIs were held with 20 HIV+ FPDs, 20 family members, 20 villagers from HIV-negative households and 20 local health workers. A further 31 participants participated in four FGDs; two each with villagers from HIV-negative households and local health workers, respectively.

Main findings

1. HIV testing and disclosure: Most of the interviewed HIV+ FPDs were tested when the local CDC went to their villages and offered testing. Most of their spouses were also tested. Villagers usually knew who is HIV+ in their village because there have been confidentiality issues in the notification process and because they see who is seeking AIDS-related healthcare or getting assistance from the government's HIV/AIDS care and support programs.
2. Discrimination and stigma: There have been no acts of physical violence as a result of discrimination or stigma. Acts of discrimination included being deliberately ignored, both by other villagers and their families. Stigma associated with HIV/AIDS includes imminent death, loss of labor and family economy, and bad reputation. The severity of stigma/discrimination is inversely related to the prevalence of HIV in a village.
3. Psychological status: The ART program has improved people's outlook on life, however many remain pessimistic about their health, economic situation and future.
4. HIV knowledge: Almost all the interviewees had heard of HIV/AIDS and knew the three main transmission routes (i.e. blood, sex, mother-to-child), however there were some misconceptions about transmission and prevention.
5. Sexual behavior: Most of the HIV+ FPDs reduced their frequency of sex, and some even stopped having sex, after they learned their sero-status. Extra-marital sex was rare. HIV+ FPDs rarely used condoms before they knew they were positive. While they reported that they now use condoms every time they have sex, some of them do not use condoms correctly.
6. Healthcare seeking behavior: After the introduction of the Four Free and One Care program, HIV+ FPDs tended to seek health services in HIV-designated hospitals/clinics because they provide financial support for medications. Despite the subsidies, many still found healthcare unaffordable. A minority forgot to take or could not adhere to their regimen at first, however this situation was very much improved by regular home visits by local health workers.
7. Social network and support: Social networks among HIV+ FPDs have been formed as a result of daily life, work and medical treatment. However the networks vary. In Funan, a stable network has been formed among HIV+ people who know each other quite well because they live close to each other and were together when selling blood, seeking medical care after being informed of their HIV+ status and participating in AIDS-related programs. In Yingzhou, PLWHAs have less contact with each other, partly because they do not have a fixed treatment place. They do, however, have some opportunities to meet and chat with each other.
8. Perceived needs: Participants were keen to learn more about HIV in general and in particular about treatment. They also desire more opportunity for communication to help them deal with the stress and pressure they experience. Family member recognized the need for some kind of intervention to help their HIV+ relatives.
9. Economic situation: HIV+ individuals are the main income earners for their household, however most are not fit enough for jobs in the cities and rely on crops as their main source of income. People in Yingzhou are generally better off than people in Funan. A large proportion of the family income is spent on healthcare for the HIV+ family member.
10. Modality of intervention: Participants' opinions on AIDS-related programs varied widely. HIV+ participants indicated their willingness to participate in any kind of AIDS-related programs. Group activities seemed to be acceptable. It was suggested that groups be divided by gender; that activities be held in a nearby or convenient location; that the intervention be scheduled during the off-season for farming; and that village leaders or doctors act as the contact persons for AIDS-related programs.

ELIGIBILITY:
Inclusion Criteria for HIV Infected Villagers:

* HIV infected
* Between 20 and 59 years of age
* Living in Funan County or Yingzhou District, Fuyang, Anhui Province, China
* Married
* Former plasma donor

Inclusion Criteria for Family Members of HIV Infected Villagers:

* HIV uninfected
* Living in Funan County or Yingzhou District, Fuyang, Anhui Province, China
* Parent, spouse, brother, sister, or child of HIV infected participant of the study
* Aware of participating family member's HIV-positive status

Inclusion Criteria for Local Health Workers:

* Doctor, nurse, or other village health worker in Funan County or Yingzhou District, Fuyang, Anhui Province, China
* Working at county or township hospital or clinic in study villages in either Funan County or Yingzhou District, Fuyang, Anhui Province, China

Inclusion Criteria for Villagers Who Are Not From Households with an HIV Infected Participant:

* HIV uninfected OR unknown HIV status
* Between 18 and 59 years of age
* Living in Funan County or Yingzhou District, Fuyang, Anhui Province, China
* Not a family member of someone who is HIV infected

Exclusion Criteria:

* Traveled outside of Funan County and Yingzhou District, Fuyang, Anhui Province, China for more than 6 months in the year prior to study entry
* Permanent disability such as deafness, serious mental illness, or mental retardation that may interfere with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected former plasma donors (FPDs) , family members of HIV-infected FPDs, local healthcare workers and villagers not related to an HIV-infected individual in Fuyang, Anhui Province, China
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2004-10; Primary Completion 2005-03 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zunyou Wu, MD, PhD, Study Chair — Division of Health Education and Behavioral Intervention, National Center for AIDS/STD Control and Prevention, Chinese Center for Disease Control and Prevention; Mary Jane Rotheram-Borus, PhD, Study Chair — Division of Social and Community Psychiatry, Neuropsychiatric Institute, University of California, Los Angeles; Jie Xu, MD, MS, MPH, Study Chair — Division of Health Education and Behavioral Intervention, National Center for AIDS/STD Control and Prevention, Chinese Center for Disease Control and Prevention

REFERENCES:
- [Background] Cao X, Sullivan SG, Xu J, Wu Z; China CIPRA Project 2 Team. Understanding HIV-related stigma and discrimination in a "blameless" population. AIDS Educ Prev. 2006 Dec;18(6):518-28. doi: 10.1521/aeap.2006.18.6.518. PMID 17166078
- [Background] Chen J, Choe MK, Chen S, Zhang S. Community environment and HIV/AIDS-related stigma in China. AIDS Educ Prev. 2005 Feb;17(1):1-11. doi: 10.1521/aeap.17.1.1.58689. PMID 15843106
- [Background] Feng G, Pang L, Wu Z. Impact of being willing to disclose HIV sero-status on voluntary counseling and testing, Chinese J AIDS/STD, 2005, 11: 237-238 (Chinese)
- [Background] Wang X, Wu Z. Factors associated with adherence to ARV among AIDS patients and related intervention, Chinese J AIDS/STD, 2005, 11, 225-227 (Chinese)
- [Background] Xu J, Sullivan SG, Dou Z, Wu Z; China CIPRA Project 2 Team. Economic stress and HIV-associated health care utilization in a rural region of China: a qualitative study. AIDS Patient Care STDS. 2007 Nov;21(11):787-98. doi: 10.1089/apc.2007.0005. PMID 17944555